CLINICAL TRIAL: NCT04259164
Title: Evaluation of the Anti-inflammatory Effects of Glycopyrronium Added to Indacaterol/Mometasone on the Allergen-induced Late Asthmatic Response
Brief Title: Anti-inflammatory Effects Glycopyrronium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Maarten van den Berge, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ABR70842
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Asthma; Allergic Asthma
Keywords: Asthma; Anti-inflammatory; Allergen
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; QMF149; indacaterol

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, two-way cross-over study with two treatment periods.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QMF149 (Active Comparator): Mometasone furoaat / Indacaterol
  Interventions: Drug: QMF149
- QVM149 (Experimental): Mometasone furoaat / Indacaterol / Glycopyrronium
  Interventions: Drug: QVM149

INTERVENTIONS:
Drug: QVM149 — Anti-inflammatory effect of Glycopyrronium added to Mometasone / Indacaterol
  Other Names: Mometasone/Indacaterol/Glycopyrronium
  Arms: QVM149
Drug: QMF149 — Mometasone / Indacaterol
  Other Names: Mometasone/Indacaterol
  Arms: QMF149

SUMMARY:
Double-blind, randomized, two-way cross-over study with two treatment periods. 28 subjects with asthma will be randomized in 1:1 ratio to treatment A) Indacaterol/Mometasone 150/160 μg once daily and treatment B) Indacaterol/Glycopyrronium/Mometasone 150/50/80 μg once daily for period 1. For period 2, subjects will be crossed over to the other treatment arm. Subjects will be screened during the first visit. After inclusion subjects will be seen for 3 visits during the Run-in period, 3 visits during treatment period 1 and 3 visits during treatment period 2. During these visits patients will be clinically characterized and exposed to allergen challenge tests.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female adult patients aged between 18 and 65 years old.
* Patients with a diagnosis of asthma for at least 6 months prior to Visit 1 with current asthma severity of step 1-3 (GINA 2018).
* Patients with presence of allergy against house dust mite, cat or grass pollen.
* PC20 histamine or equivalent ≤ 8 mg/ml.
* Drop in FEV1 > 20% during the early asthmatic response and drop in FEV1 > 15% during the late asthmatic response, i.e. between 3-8 hours after allergen challenge.
* Patients able to produce sputum of sufficient quality for evaluation of cell differential counts 24 hours after the baseline allergen challenge at Visit 3.

Exclusion Criteria:

* Smoking history ≥ 10 pack-years. Ex-smokers are eligible for inclusion if they quit smoking for at least 6 months prior to Visit 1.
* Diagnosed with Chronic Obstructive Pulmonary Disease (COPD).
* FEV1 < 70% of predicted at baseline or < 1.5 liters.
* An asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of Visit 1.
* Respiratory tract infection or clinically significant asthma worsening as defined by Investigator within 4 weeks prior to Visit 1.
* Ever required intubation for a severe asthma attack/exacerbation.
* Presence of clinical condition which is likely to be worsened by ICS administration (e.g. glaucoma, cataract and fragility fractures).
* Treated with LAMA for asthma within 3 months prior to Visit 1.
* Known with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH) or bladder-neck obstruction or severe renal impairment or urinary retention.
* Known with any chronic conditions affecting the upper respiratory tract (e.g. chronic sinusitis or polyposis nasi) which in the opinion of the investigator may interfere with the study evaluation or optimal participation in the study. Allergic rhinitis is allowed.
* History of chronic lung diseases other than asthma, including (but not limited to) sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Uncontrolled Type I or Type II diabetes.
* Clinically significant laboratory abnormality at Visit 1.
* Use of other investigational drugs within 30 days or 5 half-lives of enrollment, until the expected pharmacodynamics effect has returned to baseline, whichever is longer.
* Clinically significant condition such as (but not limited to) unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV left ventricular failure, arrhythmia, uncontrolled hypertension, cerebrovascular disease, psychiatric disease, neurodegenerative diseases, or other neurological disease, uncontrolled hypo- and hyperthyroidism and other autoimmune diseases, hypokalemia, hyper adrenergic state, or ophthalmologic disorder or patients with a medical condition that might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study.
* Diagnosis of paroxysmal (e.g., intermittent) atrial fibrillation.
* History of myocardial infarction within 12 months prior to Visit 1.
* Concomitant use of agents known to prolong the QT interval unless it can be permanently discontinued for the duration of study.
* History of long QT syndrome or QTc measured at Visit 1 (Fridericia method) is prolonged (> 450 msec for males and > 460 msec for females).
* Clinically significant ECG abnormality at Visit 1.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* History of hypersensitivity to lactose, any of the study drugs or its excipients, or to similar drugs within the class including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
* On maintenance immunotherapy (desensitization) for allergies for less than 3 months prior to Visit 1 or patients on Maintenance Immunotherapy for more than 3 months prior to Visit 1 but expected to change throughout the course of the study.
* Unable to use the Breezhaler dry powder inhaler or a metered dose inhaler.
* History of alcohol or other substance abuse that based on judgement of the investigator would interfere with study conduct.
* Known history of non-compliance to medication.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment and for 5-times the terminal half-life after stopping medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
% of sputum eosinophils | 24 hours after allergen challenge at the end of each treatment period vs. control allergen challenge
  Percentage of sputum eosinophils

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Van den Berge, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands